CLINICAL TRIAL: NCT05372575
Title: A COHORT STUDY TO EVALUATE IMMUNOGENICITY FOR CHILDREN AGED 5 MONTHS TO ≤60 MONTHS AT THE TIME OF CLINICAL PNEUMONIA DIAGNOSIS
Brief Title: A COHORT STUDY TO EVALUATE IMMUNOGENICITY FOR CHINESE CHILDREN AT THE TIME OF CLINICAL PNEUMONIA DIAGNOSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1851196; 2022-000845-34 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-05-12 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-12

CONDITIONS: Immunogenicity, Vaccine
Keywords: Serum concentrations of anticapsular immunoglobulin G (IgG) and serum levels of opsonophagocytic activity (OPA) for the PCV13 pneumococcal serotypes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCV13 group and non PCV13 group (Other): This study plan to recruit those young patients who have or not have got PCV13 vaccine before study start
  Interventions: Biological: PCV13 PAC study

INTERVENTIONS:
Biological: PCV13 PAC study — To test the serotype-specific IgG geometric mean concentration (GMC) and MOPA geometric mean titers (GMT) for each of the pneumococcal serotypes measured at the time of diagnosis of clinical pneumonia.

SUMMARY:
This is a PAC study after PCV13 launch in China. Based on recommendation from China Agency, Pfizer was required to conduct a descriptive immunogenicity study to measure the antibody levels at the time of disease onset.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the parent(s)/legal guardian has been informed of all pertinent aspects of the study.
2. Subjects whose caregiver is willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
3. A diagnosis of clinical pneumonia per SCH standard of care.
4. 5 months to ≤60 months of age at the time of consent.
5. Vaccination history (ie, vaccine book or picture of vaccine book) is available for confirmation.

Exclusion Criteria:

1. Infant or child who is a family member of:

   * Investigator site staff members directly involved in the conduct of the study;
   * Site staff members otherwise supervised by the investigator;
   * Pfizer employees directly involved in the conduct of the study.
2. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
3. Blood draw is counter indicated.
4. Previous participation in this study within 30 days.
5. Previous vaccination with licensed or investigational pneumococcal vaccine. This excludes previous vaccination with 13vPnC as per the approved recommendations in China.
6. Received blood, blood fractions, plasma, or immunoglobulins within 3 months of the study blood draw.
7. Hospital acquired pneumonia (ie, onset >48 hours after hospitalization).

Ages: 5 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Children's Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children hospitalized with a diagnosis of clinical pneumonia were considered for the study. Participants participated in the study for 1 day. Participants were followed for 12 hours after blood draw and deep respiratory aspirate if collected as a study procedure. A total of 300 participants were enrolled in this study.
Pre-assignment Details: No vaccines were administered during the study.
Groups:
- 13vPnC Cohort: The vaccination history of 13-valent pneumococcal conjugate vaccine (13vPnC) initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnc vaccination was confirmed as received, and all other inclusion/exclusion criteria were met, this participant was enrolled and assigned to the vaccinated group (ie, 13vPnC Cohort). No vaccines were administered during the study.
- Non-13vPnC Cohort: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnC vaccination was confirmed as not received, and all other inclusion / exclusion criteria were met, this participant was enrolled and assigned to the unvaccinated group (ie, Non-13vPnC Cohort). No vaccines were administered during the study.
Period: Overall Study
Arm/Group | 13vPnC Cohort | Non-13vPnC Cohort
Started | 101 | 199
Completed | 94 | 183
Not Completed | 7 | 16
Not completed — Protocol Violation | 7 | 16

BASELINE CHARACTERISTICS:
Population: Analysis population for baseline characteristics included all participants who signed the informed consent document.
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC Cohort | Non-13vPnC Cohort | Total
Number analyzed (Participants) | 101 | 199 | 300
Age, Customized [Count of Participants; unit: Participants]
  <=4 months | 1 | 0 | 1
  5-12 months | 27 | 50 | 77
  13-24 months | 39 | 49 | 88
  25-60 months | 34 | 100 | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 94 | 142
  Male | 53 | 105 | 158
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 101 | 199 | 300
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic/non-Latino | 101 | 199 | 300

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Pneumococcal Immunoglobulin G (IgG) by Cohort
Description: Approximately 5 mL of blood sample was collected within 24 hours of enrollment. Blood must have been drawn from peripheral veins (eg, arm, foot, or scalp veins). Serum concentrations of anticapsular IgG were determined by enzyme-linked immunosorbent assay (ELISA) for each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) in all participants with a collected blood sample.
Time Frame: Day 1
Population: Analysis population for this outcome measure (OM) included all participants who signed the informed consent document, met all inclusion/exclusion criteria, and had at least 1 immunogenicity assay value available for analysis. Overall number of participants analyzed indicates the number of participants in this analysis population. Number Analyzed in each row indicates the number of participants with valid and determinate assay results for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | 13vPnC Cohort | Non-13vPnC Cohort
Number analyzed (Participants) | 92 | 184
microgram per milliliter (µg/mL)
  Serotype: 1: number analyzed (Participants) | 92 | 179
  Serotype: 1 | 1.55 [1.17 to 2.06] | 0.12 [0.09 to 0.15]
  Serotype: 3 | 0.42 [0.32 to 0.54] | 0.07 [0.06 to 0.08]
  Serotype: 4 | 1.36 [1.00 to 1.84] | 0.08 [0.06 to 0.10]
  Serotype: 5 | 1.74 [1.41 to 2.15] | 0.72 [0.63 to 0.82]
  Serotype: 6A: number analyzed (Participants) | 92 | 183
  Serotype: 6A | 2.42 [1.85 to 3.15] | 0.38 [0.33 to 0.44]
  Serotype: 6B | 2.47 [1.90 to 3.22] | 0.37 [0.32 to 0.43]
  Serotype: 7F: number analyzed (Participants) | 92 | 183
  Serotype: 7F | 1.81 [1.41 to 2.32] | 0.19 [0.16 to 0.23]
  Serotype: 9V | 1.18 [0.96 to 1.46] | 0.30 [0.26 to 0.36]
  Serotype: 14: number analyzed (Participants) | 92 | 180
  Serotype: 14 | 4.67 [3.40 to 6.42] | 0.08 [0.06 to 0.10]
  Serotype: 18C: number analyzed (Participants) | 92 | 182
  Serotype: 18C | 1.03 [0.79 to 1.34] | 0.06 [0.05 to 0.08]
  Serotype: 19A | 3.19 [2.50 to 4.07] | 0.75 [0.65 to 0.86]
  Serotype: 19F: number analyzed (Participants) | 92 | 181
  Serotype: 19F | 3.31 [2.53 to 4.31] | 0.38 [0.31 to 0.46]
  Serotype: 23F | 2.04 [1.56 to 2.68] | 0.25 [0.21 to 0.28]
Statistical Analysis 1: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; Geometric mean ratio (GMR) of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 1; Test type: Superiority — The 2-sided 95% confidential interval (CI) on the GMRs (the GMC of 13vPnC Cohort to the GMC of Non-13vPnC Cohort) for all 13 serotypes are provided and those 95% CIs were constructed by back transformation of the CIs for the mean difference of the measures on the logarithmically transformed scale (IgG) using Student's t distribution; Geometric Mean Ratio (GMR) = 13.16, 95% CI 2-sided [8.99 to 19.28] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 2: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 3; Test type: Superiority — The 2-sided 95% CI on the GMRs (the GMC of 13vPnC Cohort to the GMC of Non-13vPnC Cohort) for all 13 serotypes are provided and those 95% CIs were constructed by back transformation of the CIs for the mean difference of the measures on the logarithmically transformed scale (IgG) using Student's t distribution; GMR = 5.88, 95% CI 2-sided [4.32 to 8.01] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 3: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 17.98, 95% CI 2-sided [12.07 to 26.78] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 4: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 2.42, 95% CI 2-sided [1.90 to 3.08] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 5: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 6A; Test type: Superiority — The 2-sided 95% CI on GMRs (the GMC of 13vPnC Cohort to the GMC of Non-13vPnC Cohort) for all 13 serotypes are provided and those 95% CIs were constructed by back transformation of the CIs for the mean difference of the measures on the logarithmically transformed scale (IgG) using Student's t distribution; GMR = 6.35, 95% CI 2-sided [4.68 to 8.61] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 6: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 6.64, 95% CI 2-sided [4.92 to 8.97] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 7: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 9.42, 95% CI 2-sided [6.91 to 12.83] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 8: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 3.89, 95% CI 2-sided [2.96 to 5.10] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 9: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 62.13, 95% CI 2-sided [40.16 to 96.12] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 10: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 16.37, 95% CI 2-sided [11.22 to 23.89] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 11: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 4.25, 95% CI 2-sided [3.22 to 5.62] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 12: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 8.73, 95% CI 2-sided [6.24 to 12.21] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)
Statistical Analysis 13: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 8.33, 95% CI 2-sided [6.15 to 11.29] — GMR=(GMC of 13vPnC Cohort)/(GMC of Non-13vPnC Cohort)

2. Primary Outcome: Geometric Mean Titers (GMTs) of Pneumococcal Multiplex Opsonophagocytic Activity (MOPA) by Cohort
Description: Approximately 5 mL of blood sample was collected within 24 hours of enrollment. Blood must have been drawn from peripheral veins (eg, arm, foot, or scalp veins). Serum levels of MOPA for each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all 13vPnC cohort participants with adequate blood volume. In the Non-13vPnC cohort, a sample of participants with adequate blood volume was selected, to be equal to the number of the 13vPnC Cohort included for MOPA testing. Titer was expressed as reciprocal of the highest serum dilution.
Time Frame: Day 1
Population: Analysis population for this OM included all participants who signed the informed consent document, met all inclusion/exclusion criteria, and had at least 1 immunogenicity assay value available for analysis. Overall number of participants analyzed indicates the number of participants in this analysis population. Number Analyzed in each row indicates the number of participants with valid and determinate assay results for the specified serotype.
Measure: Number (95% Confidence Interval); unit: Titers
Arm/Group | 13vPnC Cohort | Non-13vPnC Cohort
Number analyzed (Participants) | 92 | 184
Titers
  Serotype: 1: number analyzed (Participants) | 61 | 69
  Serotype: 1 | 70.9 [40.8 to 123.3] | 14.8 [9.2 to 24.0]
  Serotype: 3: number analyzed (Participants) | 61 | 69
  Serotype: 3 | 272.8 [173.9 to 428.0] | 30.1 [18.7 to 48.4]
  Serotype: 4: number analyzed (Participants) | 61 | 69
  Serotype: 4 | 1148.4 [755.0 to 1746.6] | 79.9 [38.6 to 165.3]
  Serotype: 5: number analyzed (Participants) | 61 | 69
  Serotype: 5 | 326.5 [197.8 to 538.8] | 18.1 [10.8 to 30.2]
  Serotype: 6A: number analyzed (Participants) | 61 | 69
  Serotype: 6A | 1825.9 [1077.4 to 3094.4] | 53.9 [27.0 to 107.4]
  Serotype: 6B: number analyzed (Participants) | 61 | 69
  Serotype: 6B | 844.8 [489.7 to 1457.4] | 60.1 [31.9 to 113.4]
  Serotype: 7F: number analyzed (Participants) | 61 | 69
  Serotype: 7F | 3791.4 [2495.7 to 5759.6] | 223.2 [115.8 to 430.2]
  Serotype: 9V: number analyzed (Participants) | 61 | 69
  Serotype: 9V | 919.7 [559.9 to 1510.6] | 47.6 [27.2 to 83.3]
  Serotype: 14: number analyzed (Participants) | 61 | 69
  Serotype: 14 | 1387.9 [921.8 to 2089.8] | 132.7 [66.9 to 263.1]
  Serotype: 18C: number analyzed (Participants) | 61 | 69
  Serotype: 18C | 404.2 [255.9 to 638.5] | 33.3 [19.6 to 56.7]
  Serotype: 19A: number analyzed (Participants) | 61 | 69
  Serotype: 19A | 1046.6 [620.0 to 1766.6] | 44.3 [25.1 to 77.9]
  Serotype: 19F: number analyzed (Participants) | 61 | 69
  Serotype: 19F | 554.2 [344.6 to 891.3] | 31.4 [18.5 to 53.4]
  Serotype: 23F: number analyzed (Participants) | 61 | 69
  Serotype: 23F | 3634.9 [2281.4 to 5791.3] | 81.8 [40.1 to 166.7]
Statistical Analysis 1: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 1; Test type: Superiority — The 2-sided 95% CI on the GMR (the GMT of 13vPnC Cohort to the GMT of Non-13vPnC Cohort) for all 13 serotypes are provided and those 95% CIs were constructed by back transformation of the CIs for the mean difference of the measures on the logarithmically transformed scale (MOPA) using Student's t distribution; Geometric Mean Ratio (GMR) = 4.78, 95% CI 2-sided [2.32 to 9.86] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 2: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 3; Test type: Superiority — The 2-sided 95% CI on the GMRs (the GMT of 13vPnC Cohort to the GMT of Non-13vPnC Cohort) for all 13 serotypes are provided and those 95% CIs were constructed by back transformation of the CIs for the mean difference of the measures on the logarithmically transformed scale (MOPA) using Student's t distribution; GMR = 9.06, 95% CI 2-sided [4.72 to 17.39] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 3: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 14.37, 95% CI 2-sided [6.25 to 33.05] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 4: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 18.03, 95% CI 2-sided [8.84 to 36.80] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 5: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 6A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 33.88, 95% CI 2-sided [14.33 to 80.13] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 6: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 14.05, 95% CI 2-sided [6.07 to 32.52] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 7: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 16.99, 95% CI 2-sided [7.85 to 36.76] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 8: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 19.31, 95% CI 2-sided [9.13 to 40.84] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 9: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 10.46, 95% CI 2-sided [4.74 to 23.10] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 10: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 12.13, 95% CI 2-sided [6.00 to 24.51] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 11: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 23.65, 95% CI 2-sided [10.94 to 51.10] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 12: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 17.62, 95% CI 2-sided [8.65 to 35.93] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)
Statistical Analysis 13: Comparison: 13vPnC Cohort vs Non-13vPnC Cohort; GMR of 13vPnC Cohort/Non-13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 44.46, 95% CI 2-sided [19.11 to 103.43] — GMR=(GMT of 13vPnC Cohort)/(GMT of Non-13vPnC Cohort)

3. Primary Outcome: GMCs of Pneumococcal IgG by Cohort and Vaccine Type (VT) Carriage Status - Subgroup Analysis
Description: Approximately 5 mL of blood sample was collected within 24 hours of enrollment. Blood must have been drawn from peripheral veins (eg, arm, foot, or scalp veins). Serum concentrations of anticapsular IgG were determined by ELISA for each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) in all participants with a collected blood sample. For each cohort, participants were assigned to 2 subgroups: Participant in whom a 13vPnC VT strain had been isolated from the respiratory tract, and participant from whom a 13vPnC VT strain had not been isolated from the respiratory tract (VT carrier versus without VT carrier).
Time Frame: Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Groups:
- 13vPnC Cohort: VT+ Subgroup: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnc vaccination was confirmed as received, and all other inclusion/exclusion criteria were met, this participant was enrolled and assigned to the vaccinated group (ie, 13vPnC Cohort). Participants in this subgroup had a 13vPnC VT strain isolated from the respiratory tract (VT+). No vaccines were administered during the study.
- 13vPnC Cohort: VT- or Sp- Subgroup: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnc vaccination was confirmed as received, and all other inclusion/exclusion criteria were met, this participant was enrolled and assigned to the vaccinated group (ie, 13vPnC Cohort). Participants in this subgroup had no 13vPnC VT strain isolated from the respiratory tract (VT-) or had negative S. pneumoniae (Sp-). No vaccines were administered during the study.
- Non-13vPnC Cohort: VT+ Subgroup: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnC vaccination was confirmed as not received, and all other inclusion / exclusion criteria were met, this participant was enrolled and assigned to the unvaccinated group (ie, Non-13vPnC Cohort). Participants in this subgroup had a 13vPnC VT strain isolated from the respiratory tract (VT+). No vaccines were administered during the study.
- Non-13vPnC Cohort: VT- or Sp- Subgroup: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnC vaccination was confirmed as not received, and all other inclusion / exclusion criteria were met, this participant was enrolled and assigned to the unvaccinated group (ie, Non-13vPnC Cohort). Participants in this subgroup had no 13vPnC VT strain isolated from the respiratory tract (VT-) or had negative S. pneumoniae (Sp-). No vaccines were administered during the study.
Arm/Group | 13vPnC Cohort: VT+ Subgroup | 13vPnC Cohort: VT- or Sp- Subgroup | Non-13vPnC Cohort: VT+ Subgroup | Non-13vPnC Cohort: VT- or Sp- Subgroup
Number analyzed (Participants) | 7 | 79 | 20 | 140
microgram per milliliter (µg/mL)
  Serotype: 1: number analyzed (Participants) | 7 | 79 | 20 | 136
  Serotype: 1 | 0.81 [0.28 to 2.33] | 1.69 [1.23 to 2.31] | 0.08 [0.04 to 0.18] | 0.12 [0.09 to 0.16]
  Serotype: 3 | 0.32 [0.10 to 1.04] | 0.44 [0.33 to 0.58] | 0.05 [0.03 to 0.09] | 0.07 [0.06 to 0.09]
  Serotype: 4 | 0.97 [0.26 to 3.64] | 1.43 [1.02 to 2.00] | 0.05 [0.02 to 0.11] | 0.07 [0.05 to 0.09]
  Serotype: 5 | 1.45 [0.51 to 4.15] | 1.77 [1.41 to 2.24] | 0.58 [0.40 to 0.83] | 0.72 [0.61 to 0.85]
  Serotype: 6A | 1.78 [0.73 to 4.32] | 2.59 [1.93 to 3.48] | 0.34 [0.22 to 0.51] | 0.36 [0.31 to 0.43]
  Serotype: 6B | 1.94 [0.78 to 4.81] | 2.60 [1.93 to 3.50] | 0.51 [0.31 to 0.84] | 0.33 [0.28 to 0.40]
  Serotype: 7F: number analyzed (Participants) | 7 | 79 | 20 | 139
  Serotype: 7F | 0.83 [0.36 to 1.92] | 1.97 [1.50 to 2.59] | 0.14 [0.07 to 0.29] | 0.19 [0.15 to 0.23]
  Serotype: 9V | 0.97 [0.37 to 2.53] | 1.21 [0.96 to 1.54] | 0.22 [0.10 to 0.46] | 0.30 [0.25 to 0.36]
  Serotype: 14: number analyzed (Participants) | 7 | 79 | 19 | 138
  Serotype: 14 | 3.29 [0.49 to 21.91] | 4.96 [3.54 to 6.94] | 0.04 [0.02 to 0.09] | 0.08 [0.06 to 0.12]
  Serotype: 18C: number analyzed (Participants) | 7 | 79 | 20 | 138
  Serotype: 18C | 0.65 [0.30 to 1.44] | 1.08 [0.81 to 1.45] | 0.04 [0.02 to 0.09] | 0.06 [0.05 to 0.08]
  Serotype: 19A | 4.69 [2.35 to 9.38] | 3.02 [2.30 to 3.97] | 0.58 [0.37 to 0.90] | 0.74 [0.63 to 0.86]
  Serotype: 19F: number analyzed (Participants) | 7 | 79 | 20 | 138
  Serotype: 19F | 5.80 [1.41 to 23.82] | 3.22 [2.41 to 4.28] | 0.38 [0.21 to 0.68] | 0.33 [0.26 to 0.42]
  Serotype: 23F | 1.04 [0.47 to 2.32] | 2.23 [1.65 to 3.02] | 0.25 [0.15 to 0.40] | 0.23 [0.20 to 0.27]
Statistical Analysis 1: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 1; Test type: Superiority — [test comment as in outcome 1, analysis 2]; Geometric Mean Ratio (GMR) = 0.48, 95% CI 2-sided [0.16 to 1.42] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 2: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 3; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.74, 95% CI 2-sided [0.27 to 1.98] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 3: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.68, 95% CI 2-sided [0.21 to 2.19] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 4: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.82, 95% CI 2-sided [0.36 to 1.86] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 5: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 6A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.68, 95% CI 2-sided [0.25 to 1.89] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 6: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.74, 95% CI 2-sided [0.27 to 2.07] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 7: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.42, 95% CI 2-sided [0.16 to 1.09] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 8: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.80, 95% CI 2-sided [0.35 to 1.81] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 9: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.66, 95% CI 2-sided [0.20 to 2.24] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 10: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.60, 95% CI 2-sided [0.22 to 1.65] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 11: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 1.55, 95% CI 2-sided [0.61 to 3.93] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 12: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 1.80, 95% CI 2-sided [0.65 to 4.99] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 13: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.47, 95% CI 2-sided [0.17 to 1.31] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 14: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 1; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.65, 95% CI 2-sided [0.31 to 1.38] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 15: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 3; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.70, 95% CI 2-sided [0.40 to 1.24] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 16: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.73, 95% CI 2-sided [0.33 to 1.59] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 17: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.80, 95% CI 2-sided [0.52 to 1.25] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 18: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 6A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.93, 95% CI 2-sided [0.57 to 1.52] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 19: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 1.53, 95% CI 2-sided [0.95 to 2.47] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 20: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.74, 95% CI 2-sided [0.41 to 1.34] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 21: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.73, 95% CI 2-sided [0.34 to 1.57] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 22: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.44, 95% CI 2-sided [0.16 to 1.18] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 23: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.59, 95% CI 2-sided [0.25 to 1.40] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 24: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 0.79, 95% CI 2-sided [0.50 to 1.23] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 25: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 1.14, 95% CI 2-sided [0.60 to 2.18] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 26: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 1.08, 95% CI 2-sided [0.68 to 1.72] — GMR=(GMC of VT+ Subgroup)/(GMC of VT- or Sp- Subgroup)
Statistical Analysis 27: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 1; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 10.30, 95% CI 2-sided [2.44 to 43.49] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 28: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 3; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 6.17, 95% CI 2-sided [2.07 to 18.42] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 29: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 4; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 18.70, 95% CI 2-sided [4.35 to 80.37] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 30: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 2.50, 95% CI 2-sided [1.14 to 5.52] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 31: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 6A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 5.24, 95% CI 2-sided [2.33 to 11.80] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 32: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 6B; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 3.77, 95% CI 2-sided [1.47 to 9.65] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 33: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 7F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 5.94, 95% CI 2-sided [1.65 to 21.36] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 34: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 9V; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 4.44, 95% CI 2-sided [1.17 to 16.87] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 35: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 14; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 90.80, 95% CI 2-sided [16.67 to 494.56] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 36: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 18C; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 17.83, 95% CI 2-sided [3.79 to 83.78] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 37: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 19A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 8.11, 95% CI 2-sided [3.60 to 18.30] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 38: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 19F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 15.29, 95% CI 2-sided [4.64 to 50.35] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 39: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 23F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 4.19, 95% CI 2-sided [1.72 to 10.25] — GMR=(GMC of 13vPnC VT+ Subgroup)/(GMC of non-13vPnC VT+ Subgroup)
Statistical Analysis 40: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 1; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 13.93, 95% CI 2-sided [9.14 to 21.23] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 41: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 3; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 5.86, 95% CI 2-sided [4.17 to 8.24] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 42: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 4; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 19.97, 95% CI 2-sided [12.80 to 31.15] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 43: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 5; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 2.46, 95% CI 2-sided [1.87 to 3.24] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 44: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 6A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 7.12, 95% CI 2-sided [5.05 to 10.03] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 45: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 6B; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 7.78, 95% CI 2-sided [5.54 to 10.92] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 46: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 7F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 10.40, 95% CI 2-sided [7.40 to 14.61] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 47: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 9V; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 4.07, 95% CI 2-sided [3.04 to 5.47] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 48: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 14; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 60.32, 95% CI 2-sided [37.25 to 97.67] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 49: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 18C; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 17.35, 95% CI 2-sided [11.37 to 26.47] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 50: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 19A; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 4.11, 95% CI 2-sided [3.00 to 5.62] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 51: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 19F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 9.68, 95% CI 2-sided [6.65 to 14.08] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 52: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 23F; Test type: Superiority — [test comment as in outcome 1, analysis 2]; GMR = 9.70, 95% CI 2-sided [6.90 to 13.64] — GMR=(GMC of 13vPnC VT- or Sp- Subgroup)/(GMC of non-13vPnC VT- or Sp- Subgroup)

4. Primary Outcome: GMTs of Pneumococcal MOPA by Cohort and VT Carriage Status - Subgroup Analysis
Description: Approximately 5 mL of blood sample was collected within 24 hours of enrollment. Blood must have been drawn from peripheral veins (eg, arm, foot, or scalp veins). Serum levels of MOPA for each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all 13vPnC cohort participants with adequate blood volume. In the Non-13vPnC cohort, a sample of participants with adequate blood volume was selected, to be equal to the number of the 13vPnC Cohort included for MOPA testing. For each cohort, participants were assigned to 2 subgroups: Participant in whom a 13vPnC VT strain had been isolated from the respiratory tract, and participant from whom a 13vPnC VT strain had not been isolated from the respiratory tract (VT carrier versus without VT carrier). Titer was expressed as reciprocal of the highest serum dilution.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Titers
Groups:
- Non-13vPnC Cohort: VT- or Sp- Subgroup: The vaccination history of 13vPnC initially was obtained either from the participant's parent/caregiver; confirmation of 13vPnC receipt from vaccine book or image of vaccine book was required. If 13vPnC vaccination was confirmed as not received, and all other inclusion / exclusion criteria were met, this participant was enrolled and assigned to the unvaccinated group (Non-13vPnC Cohort). Participants in this subgroup had no 13vPnC VT strain isolated from the respiratory tract (VT-) or had negative S. pneumoniae (Sp-). No vaccines were administered during the study.
Arm/Group | 13vPnC Cohort: VT+ Subgroup | 13vPnC Cohort: VT- or Sp- Subgroup | Non-13vPnC Cohort: VT+ Subgroup | Non-13vPnC Cohort: VT- or Sp- Subgroup
Number analyzed (Participants) | 7 | 79 | 20 | 140
Titers
  Serotype: 1: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 1 | 35.0 [2.2 to 547.7] | 71.1 [38.4 to 131.4] | 11.1 [4.1 to 30.5] | 14.6 [8.4 to 25.4]
  Serotype: 3: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 3 | 146.6 [35.6 to 602.7] | 273.7 [163.5 to 458.2] | 29.2 [14.0 to 61.0] | 28.6 [16.3 to 50.1]
  Serotype: 4: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 4 | 522.0 [165.0 to 1651.2] | 1154.4 [726.1 to 1835.4] | 38.1 [6.7 to 216.9] | 86.1 [37.4 to 198.3]
  Serotype: 5: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 5 | 539.5 [41.4 to 7035.5] | 302.7 [173.2 to 529.0] | 11.1 [3.6 to 34.7] | 17.6 [9.9 to 31.4]
  Serotype: 6A: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 6A | 482.4 [31.8 to 7306.4] | 2110.3 [1176.4 to 3785.6] | 46.1 [5.8 to 366.1] | 52.5 [23.7 to 116.2]
  Serotype: 6B: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 6B | 69.4 [1.4 to 3480.8] | 1099.1 [639.5 to 1889.0] | 102.7 [14.2 to 742.0] | 53.9 [26.4 to 110.3]
  Serotype: 7F: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 7F | 4661.3 [2222.1 to 9777.9] | 3837.7 [2367.8 to 6220.2] | 442.5 [87.9 to 2228.3] | 180.8 [84.0 to 389.4]
  Serotype: 9V: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 9V | 215.9 [6.7 to 6985.7] | 1074.9 [637.7 to 1811.9] | 65.0 [13.3 to 318.0] | 45.3 [23.7 to 86.6]
  Serotype: 14: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 14 | 578.9 [89.2 to 3755.8] | 1617.3 [1046.6 to 2499.2] | 289.1 [22.7 to 3682.3] | 125.9 [59.7 to 265.4]
  Serotype: 18C: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 18C | 364.1 [83.5 to 1587.8] | 443.2 [265.2 to 740.7] | 22.3 [5.3 to 93.2] | 34.4 [19.2 to 61.8]
  Serotype: 19A: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 19A | 1515.6 [296.4 to 7750.1] | 1122.7 [622.0 to 2026.5] | 62.7 [8.6 to 456.6] | 41.6 [22.1 to 78.3]
  Serotype: 19F: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 19F | 1830.0 [240.5 to 13924.9] | 472.7 [279.4 to 799.7] | 19.3 [5.5 to 67.5] | 30.4 [16.6 to 55.7]
  Serotype: 23F: number analyzed (Participants) | 5 | 52 | 9 | 54
  Serotype: 23F | 1092.5 [140.0 to 8523.4] | 4111.0 [2442.0 to 6920.7] | 104.1 [14.5 to 746.9] | 84.4 [37.3 to 190.9]
Statistical Analysis 1: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 1; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.49, 95% CI 2-sided [0.06 to 3.91] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 2: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 3; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.54, 95% CI 2-sided [0.10 to 2.92] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 3: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.45, 95% CI 2-sided [0.10 to 2.07] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 4: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.78, 95% CI 2-sided [0.27 to 11.75] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 5: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 6A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.23, 95% CI 2-sided [0.03 to 1.65] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 6: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.06, 95% CI 2-sided [0.01 to 0.44] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 7: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.21, 95% CI 2-sided [0.56 to 2.65] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 8: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.20, 95% CI 2-sided [0.03 to 1.26] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 9: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.36, 95% CI 2-sided [0.08 to 1.55] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 10: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.82, 95% CI 2-sided [0.15 to 4.47] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 11: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.35, 95% CI 2-sided [0.19 to 9.44] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 12: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 3.87, 95% CI 2-sided [0.67 to 22.42] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 13: Comparison: 13vPnC Cohort: VT+ Subgroup vs 13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in 13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.27, 95% CI 2-sided [0.05 to 1.52] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 14: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 1; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.76, 95% CI 2-sided [0.19 to 3.07] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 15: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 3; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.02, 95% CI 2-sided [0.42 to 2.46] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 16: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 4; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.44, 95% CI 2-sided [0.05 to 3.73] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 17: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 5; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.63, 95% CI 2-sided [0.15 to 2.73] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 18: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 6A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.88, 95% CI 2-sided [0.11 to 6.99] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 19: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 6B; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.90, 95% CI 2-sided [0.29 to 12.51] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 20: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 7F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 2.45, 95% CI 2-sided [0.34 to 17.43] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 21: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 9V; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.43, 95% CI 2-sided [0.27 to 7.70] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 22: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 2.30, 95% CI 2-sided [0.30 to 17.41] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 23: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 18C; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.65, 95% CI 2-sided [0.14 to 2.97] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 24: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 19A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.51, 95% CI 2-sided [0.28 to 8.21] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 25: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 19F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.63, 95% CI 2-sided [0.13 to 2.97] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 26: Comparison: Non-13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of VT+ Subgroup/VT- or Sp- Subgroup in non-13vPnC Cohort for Serotype: 23F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 1.23, 95% CI 2-sided [0.15 to 10.24] — GMR=(GMT of VT+ Subgroup)/(GMT of VT- or Sp- Subgroup)
Statistical Analysis 27: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 1; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 3.15, 95% CI 2-sided [0.41 to 23.91] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 28: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 3; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 5.02, 95% CI 2-sided [1.45 to 17.39] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 29: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 4; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 13.70, 95% CI 2-sided [1.32 to 141.81] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 30: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 5; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 48.41, 95% CI 2-sided [6.16 to 380.54] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 31: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 6A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 10.47, 95% CI 2-sided [0.48 to 229.10] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 32: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 6B; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 0.68, 95% CI 2-sided [0.02 to 19.83] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 33: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 7F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 10.53, 95% CI 2-sided [1.98 to 55.96] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 34: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 9V; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 3.32, 95% CI 2-sided [0.19 to 56.82] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 35: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 2.00, 95% CI 2-sided [0.06 to 63.12] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 36: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 18C; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 16.31, 95% CI 2-sided [2.15 to 123.48] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 37: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 19A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 24.16, 95% CI 2-sided [1.59 to 367.81] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 38: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 19F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 95.06, 95% CI 2-sided [13.08 to 691.01] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 39: Comparison: 13vPnC Cohort: VT+ Subgroup vs Non-13vPnC Cohort: VT+ Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT+ Subgroups for Serotype: 23F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 10.49, 95% CI 2-sided [0.64 to 171.84] — GMR=(GMT of 13vPnC VT+ Subgroup)/(GMT of non-13vPnC VT+ Subgroup)
Statistical Analysis 40: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 1; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 4.86, 95% CI 2-sided [2.15 to 10.96] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 41: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 3; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 9.57, 95% CI 2-sided [4.50 to 20.36] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 42: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 4; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 13.40, 95% CI 2-sided [5.20 to 34.51] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 43: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 5; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 17.15, 95% CI 2-sided [7.76 to 37.91] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 44: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 6A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 40.20, 95% CI 2-sided [15.16 to 106.65] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 45: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 6B; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 20.38, 95% CI 2-sided [8.39 to 49.51] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 46: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 7F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 21.22, 95% CI 2-sided [8.65 to 52.07] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 47: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 9V; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 23.73, 95% CI 2-sided [10.39 to 54.19] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 48: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 14; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 12.84, 95% CI 2-sided [5.46 to 30.22] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 49: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 18C; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 12.88, 95% CI 2-sided [5.95 to 27.88] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 50: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 19A; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 26.99, 95% CI 2-sided [11.46 to 63.58] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 51: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 19F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 15.53, 95% CI 2-sided [7.02 to 34.38] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)
Statistical Analysis 52: Comparison: 13vPnC Cohort: VT- or Sp- Subgroup vs Non-13vPnC Cohort: VT- or Sp- Subgroup; GMR of 13vPnC Cohort/non-13vPnC Cohort in VT- or Sp- Subgroups for Serotype: 23F; Test type: Superiority — [test comment as in outcome 2, analysis 2]; GMR = 48.73, 95% CI 2-sided [18.67 to 127.16] — GMR=(GMT of 13vPnC VT- or Sp- Subgroup)/(GMT of non-13vPnC VT- or Sp- Subgroup)

ADVERSE EVENTS:
Time Frame: From the time of the blood draw or aspirate collection through and including 12 hours on Day 1
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | 13vPnC Cohort | Non-13vPnC Cohort
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/199
Other Adverse Events (participants affected / at risk) | 0/101 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT05372575/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT05372575/SAP_001.pdf